CLINICAL TRIAL: NCT02835859
Title: Intestinal Sweet Taste Receptor Function and Adaptation to Dietary Sugars and Sweeteners
Acronym: ISTAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Collaborators: Sanford-Burnham Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TRIMD FH 607060
Record Dates: First submitted 2016-07-12; First posted 2016-07-18 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Diabetes
Keywords: Obesity, sweet taste receptors
MeSH Terms: conditions — Diabetes Mellitus; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Group 1- Oral solution (Experimental): Participants will be randomly assigned to drink two oral solutions made of different combinations of saccharin, lactisole, acetaminophen, 3-O-methyl glucose, or glucose.
  Interventions: Other: Dietary: saccharin; Other: Estimate glucose absorptions

INTERVENTIONS:
Other: Dietary: saccharin — Assess the glycemic and hormonal responses to an oral glucose load preceded by an oral solution of NCASs (saccharin).
Other: Estimate glucose absorptions — Indirectly estimate the rate of glucose absorption and gastric emptying by using 3-O-methyglucose (3-OMG) and acetaminophen, respectively.

SUMMARY:
The purpose of this study is to collect data that will help researchers better understand the various causes of obesity and diabetes; particularly to understand how consumption of NCASs affects the way the body uses nutrients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years inclusive;
2. Men and women;
3. Able to provide written, informed consent;
4. Weight stable (± 3 kg) during the 3 months prior to enrollment;
5. BMI ≤ 25 kg/m2

Exclusion Criteria:

1. Diagnosed with any of the following co-morbidities: a) coronary artery disease, angina or heart failure, b) diabetes, c) bleeding disorders, d) infections, e) hepatitis and/or cirrhosis, f) severe asthma or chronic obstructive pulmonary disorder, g) renal insufficiency, h) bariatric surgery, i) inflammatory bowel disease or malabsorption, j) cancer within the last 3 years (except non-melanoma skin cancer or treated cervical carcinoma in situ), k) psychiatric or eating disorders, l) untreated or inadequately controlled thyroid or other endocrine disorders, m) active rheumatoid arthritis or other inflammatory rheumatic disorder;
2. Consumption of more than a can of diet beverage or a spoonful of non-caloric artificial sweeteners weekly (or each equivalent from foods) during the past month.
3. Pregnant or nursing women;
4. Current smokers (smoking within the past 3 months);
5. Known hypersensitivity to saccharin, lactisole, and acetaminophen or any of its exipients;
6. History of difficult blood sample collections or unfavorable anatomy of venous access;
7. Use of medications: a) nitrates, b) beta-blockers, c) digoxin, d) anti-diabetic agents, e) oral, injected or chronic topical steroids (inhaled steroids for mild asthma are acceptable), f) chronic use of aspirin or other non-steroidal anti-inflammatory drugs, g) other drugs known to affect immune or metabolic function and h) orlistat, phentermine or other weight loss or anorectic agents.
8. Blood pressure greater than or equal to 160/100 or less than or equal to 100/50 at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-08; Primary Completion 2016-01 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Measure in glucose concentrations | Measure over a 180 minute on Days 10, 15, 20, 25
  Glucose concentrations will be measured by the glucose oxidase method (YSI 2300 automated analyzer) and insulin, C-peptide, GLP-1 and GLP-2 concentrations by immunoassay (Mesoscale Discovery Sector Imager 2400).

CONTACTS AND LOCATIONS:
Overall Officials: George Kyriazis, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swithers SE. Artificial sweeteners produce the counterintuitive effect of inducing metabolic derangements. Trends Endocrinol Metab. 2013 Sep;24(9):431-41. doi: 10.1016/j.tem.2013.05.005. Epub 2013 Jul 10. PMID 23850261
- [Background] Kyriazis GA, Soundarapandian MM, Tyrberg B. Sweet taste receptor signaling in beta cells mediates fructose-induced potentiation of glucose-stimulated insulin secretion. Proc Natl Acad Sci U S A. 2012 Feb 21;109(8):E524-32. doi: 10.1073/pnas.1115183109. Epub 2012 Feb 6. PMID 22315413
- [Background] Nakagawa Y, Nagasawa M, Yamada S, Hara A, Mogami H, Nikolaev VO, Lohse MJ, Shigemura N, Ninomiya Y, Kojima I. Sweet taste receptor expressed in pancreatic beta-cells activates the calcium and cyclic AMP signaling systems and stimulates insulin secretion. PLoS One. 2009;4(4):e5106. doi: 10.1371/journal.pone.0005106. Epub 2009 Apr 8. PMID 19352508
- [Background] Masubuchi Y, Nakagawa Y, Ma J, Sasaki T, Kitamura T, Yamamoto Y, Kurose H, Kojima I, Shibata H. A novel regulatory function of sweet taste-sensing receptor in adipogenic differentiation of 3T3-L1 cells. PLoS One. 2013;8(1):e54500. doi: 10.1371/journal.pone.0054500. Epub 2013 Jan 15. PMID 23336004
- [Background] Simon BR, Parlee SD, Learman BS, Mori H, Scheller EL, Cawthorn WP, Ning X, Gallagher K, Tyrberg B, Assadi-Porter FM, Evans CR, MacDougald OA. Artificial sweeteners stimulate adipogenesis and suppress lipolysis independently of sweet taste receptors. J Biol Chem. 2013 Nov 8;288(45):32475-32489. doi: 10.1074/jbc.M113.514034. Epub 2013 Sep 24. PMID 24068707
- [Background] Margolskee RF, Dyer J, Kokrashvili Z, Salmon KS, Ilegems E, Daly K, Maillet EL, Ninomiya Y, Mosinger B, Shirazi-Beechey SP. T1R3 and gustducin in gut sense sugars to regulate expression of Na+-glucose cotransporter 1. Proc Natl Acad Sci U S A. 2007 Sep 18;104(38):15075-80. doi: 10.1073/pnas.0706678104. Epub 2007 Aug 27. PMID 17724332
- [Background] Dyer J, Salmon KS, Zibrik L, Shirazi-Beechey SP. Expression of sweet taste receptors of the T1R family in the intestinal tract and enteroendocrine cells. Biochem Soc Trans. 2005 Feb;33(Pt 1):302-5. doi: 10.1042/BST0330302. PMID 15667333
- [Background] Jang HJ, Kokrashvili Z, Theodorakis MJ, Carlson OD, Kim BJ, Zhou J, Kim HH, Xu X, Chan SL, Juhaszova M, Bernier M, Mosinger B, Margolskee RF, Egan JM. Gut-expressed gustducin and taste receptors regulate secretion of glucagon-like peptide-1. Proc Natl Acad Sci U S A. 2007 Sep 18;104(38):15069-74. doi: 10.1073/pnas.0706890104. Epub 2007 Aug 27. PMID 17724330
- [Background] Mace OJ, Affleck J, Patel N, Kellett GL. Sweet taste receptors in rat small intestine stimulate glucose absorption through apical GLUT2. J Physiol. 2007 Jul 1;582(Pt 1):379-92. doi: 10.1113/jphysiol.2007.130906. Epub 2007 May 10. PMID 17495045
- [Background] Fujita Y, Wideman RD, Speck M, Asadi A, King DS, Webber TD, Haneda M, Kieffer TJ. Incretin release from gut is acutely enhanced by sugar but not by sweeteners in vivo. Am J Physiol Endocrinol Metab. 2009 Mar;296(3):E473-9. doi: 10.1152/ajpendo.90636.2008. Epub 2008 Dec 23. PMID 19106249
- [Background] Ma J, Bellon M, Wishart JM, Young R, Blackshaw LA, Jones KL, Horowitz M, Rayner CK. Effect of the artificial sweetener, sucralose, on gastric emptying and incretin hormone release in healthy subjects. Am J Physiol Gastrointest Liver Physiol. 2009 Apr;296(4):G735-9. doi: 10.1152/ajpgi.90708.2008. Epub 2009 Feb 12. PMID 19221011
- [Background] Brown AW, Bohan Brown MM, Onken KL, Beitz DC. Short-term consumption of sucralose, a nonnutritive sweetener, is similar to water with regard to select markers of hunger signaling and short-term glucose homeostasis in women. Nutr Res. 2011 Dec;31(12):882-8. doi: 10.1016/j.nutres.2011.10.004. PMID 22153513
- [Background] Steinert RE, Frey F, Topfer A, Drewe J, Beglinger C. Effects of carbohydrate sugars and artificial sweeteners on appetite and the secretion of gastrointestinal satiety peptides. Br J Nutr. 2011 May;105(9):1320-8. doi: 10.1017/S000711451000512X. Epub 2011 Jan 24. PMID 21255472
- [Background] Brown RJ, Walter M, Rother KI. Ingestion of diet soda before a glucose load augments glucagon-like peptide-1 secretion. Diabetes Care. 2009 Dec;32(12):2184-6. doi: 10.2337/dc09-1185. Epub 2009 Oct 6. PMID 19808921
- [Background] Pepino MY, Klein S. Response to comment on Pepino et al. Sucralose affects glycemic and hormonal responses to an oral glucose load. Diabetes care 2013;36:2530-2535. Diabetes Care. 2014 Jun;37(6):e149. doi: 10.2337/dc14-0268. No abstract available. PMID 24855177
- [Background] Brown RJ, Walter M, Rother KI. Effects of diet soda on gut hormones in youths with diabetes. Diabetes Care. 2012 May;35(5):959-64. doi: 10.2337/dc11-2424. Epub 2012 Mar 12. PMID 22410815
- [Background] Gerspach AC, Steinert RE, Schonenberger L, Graber-Maier A, Beglinger C. The role of the gut sweet taste receptor in regulating GLP-1, PYY, and CCK release in humans. Am J Physiol Endocrinol Metab. 2011 Aug;301(2):E317-25. doi: 10.1152/ajpendo.00077.2011. Epub 2011 May 3. PMID 21540445
- [Background] Steinert RE, Gerspach AC, Gutmann H, Asarian L, Drewe J, Beglinger C. The functional involvement of gut-expressed sweet taste receptors in glucose-stimulated secretion of glucagon-like peptide-1 (GLP-1) and peptide YY (PYY). Clin Nutr. 2011 Aug;30(4):524-32. doi: 10.1016/j.clnu.2011.01.007. Epub 2011 Feb 15. PMID 21324568
- [Background] Chaikomin R, Doran S, Jones KL, Feinle-Bisset C, O'Donovan D, Rayner CK, Horowitz M. Initially more rapid small intestinal glucose delivery increases plasma insulin, GIP, and GLP-1 but does not improve overall glycemia in healthy subjects. Am J Physiol Endocrinol Metab. 2005 Sep;289(3):E504-7. doi: 10.1152/ajpendo.00099.2005. Epub 2005 May 10. PMID 15886226
- [Background] Little TJ, Pilichiewicz AN, Russo A, Phillips L, Jones KL, Nauck MA, Wishart J, Horowitz M, Feinle-Bisset C. Effects of intravenous glucagon-like peptide-1 on gastric emptying and intragastric distribution in healthy subjects: relationships with postprandial glycemic and insulinemic responses. J Clin Endocrinol Metab. 2006 May;91(5):1916-23. doi: 10.1210/jc.2005-2220. Epub 2006 Feb 21. PMID 16492694
- [Background] Shirazi-Beechey SP, Moran AW, Batchelor DJ, Daly K, Al-Rammahi M. Glucose sensing and signalling; regulation of intestinal glucose transport. Proc Nutr Soc. 2011 May;70(2):185-93. doi: 10.1017/S0029665111000103. Epub 2011 Mar 30. PMID 21450125
- [Background] Ma J, Chang J, Checklin HL, Young RL, Jones KL, Horowitz M, Rayner CK. Effect of the artificial sweetener, sucralose, on small intestinal glucose absorption in healthy human subjects. Br J Nutr. 2010 Sep;104(6):803-6. doi: 10.1017/S0007114510001327. Epub 2010 Apr 27. PMID 20420761
- [Background] Jiang P, Cui M, Zhao B, Liu Z, Snyder LA, Benard LM, Osman R, Margolskee RF, Max M. Lactisole interacts with the transmembrane domains of human T1R3 to inhibit sweet taste. J Biol Chem. 2005 Apr 15;280(15):15238-46. doi: 10.1074/jbc.M414287200. Epub 2005 Jan 24. PMID 15668251
- [Background] Saccharin and its salts. IARC Monogr Eval Carcinog Risks Hum. 1999;73:517-624. No abstract available. PMID 10804968
- [Derived] Karimian Azari E, Smith KR, Yi F, Osborne TF, Bizzotto R, Mari A, Pratley RE, Kyriazis GA. Inhibition of sweet chemosensory receptors alters insulin responses during glucose ingestion in healthy adults: a randomized crossover interventional study. Am J Clin Nutr. 2017 Apr;105(4):1001-1009. doi: 10.3945/ajcn.116.146001. Epub 2017 Mar 1. PMID 28251932
- See also: Florida Hospital Translational Research Institute for Metabolism and Diabetes — http://www.tri-md.org